CLINICAL TRIAL: NCT01918839
Title: Clinical Study to Evaluate the Efficacy and Safety of Injection With VINCI Plus as Compared to Restylane-L in Correction of Nasolabial Fold
Brief Title: Efficacy and Safety of Injection With VINCI Plus Hyaluronic Acid Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D.med (Industry)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMEDVINCI001; DMEDVINCI001 (Other: D. Med)
Record Dates: First submitted 2013-08-02; First posted 2013-08-08 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Nasolabial Fold Improvement
Keywords: Investigational Device (VINCI Plus); Correction of nasolabial fold; Wrinkle improvement; Wrinkle correction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VINCI Plus (Experimental): One side has been treated with VINCI Plus
  Interventions: Device: VINCI Plus
- Restylane-L (Active Comparator): One side has been treated with Restylane-L
  Interventions: Device: Restylane-L

INTERVENTIONS:
Device: VINCI Plus — VINCI Plus 1ml injected into wrinkle treatment area
  Arms: VINCI Plus
Device: Restylane-L — Restylane-L injected into wrinkle treatment area
  Arms: Restylane-L

SUMMARY:
This clinical trial is intended to evaluate the efficacy and safety of injection with VINCI Plus as compared to Restylane-L® in correction of nasolabial fold.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 30-65, at the point of screening, wrinkles on both sides of treatment area (nasolabial fold) are in the 3rd or 4th level on the WSRS(Wrinkle Severity Rating Score)
* Surrounding soft tissue of wrinkles on both sides of nose and lips are sagging
* Wrinkles of both sides of nose and lips are visually symmetric
* Agrees to stop all other treatment of facial wrinkle improvement including dermatology treatment during clinical trial
* Able to understand and follow instructions and participate the entire period of the clinical trial
* Subject voluntarily agrees to participate in clinical trial and gives informed written consent

Exclusion Criteria:

* At the point of screening, intradermal test results show skin irritation to medical devices of clinical trial
* Within 2 weeks before the date of screening, subject has taken antithrombotic (with the exception of low dose aspirin 100mg, up to 300mg/day) or non-steroidal anti-inflammatory medication
* Case where subject has abnormal liver function or blood coagulation, has to take antithrombotic medication (with the exception of low dose aspirin 100mg, up to 300mg/day) during clinical trial
* Subject has used facial topical liniment (steroids, retinoids: excluding only medicines and cosmetics) within 4 weeks before date of screening or plans to continue using facial topical liniment during clinical trial
* Within 6 months before date of screening, subject has received anti-wrinkle or acne treatment
* Within 6 months before date of screening, subject has received facial microdermabrasion treatment, skin regeneration/rejuvenation treatment, plastic surgery, or cosmetic surgery (including Botox injections)
* Within 1 year before date of screening, subject has received CaHA (Calcium Hydroxyapatite) treatment on clinical trial medical device treatment area
* Subject has cured facial gel (Softform) or silicone implants inserted as permanent facial expansion
* Within 1 year before, subject had an illness that caused scarring or has scars on clinical trial medical device treatment area
* Subject has facial skin disease or skin wound infection that affects the clinical trial
* Weak immune system or suspect that the immune system is weak
* History of anaphylaxis or severe allergic complexity
* History of hypertrophic scar or keloid
* In the past, if there were adverse effects from EMLA Cream (if EMLA Cream was not used, the exclusion criteria for subjects applicable)
* History of hypersensitivity to Lidocaine
* Cardiovascular, digestive, respiratory, endocrine, central nervous system disorders that seems clinically significant or had a mental illness that had a significant impact on a previous clinical trial or currently has a mental illness
* Within 30 days before screening, subject participated in other clinical trials
* Female subjects of childbearing potential does not agree to a medically accepted method of contraception for the period of the clinical trial Medically acceptable methods of contraception: condoms; oral contraception continued for at least three months; or if intrauterine is used, installed a contraceptive device
* Pregnant women or nursing mothers
* In addition to the above, the test director or person in charge medically judges there are clinically significant findings that are improper for the clinical trial

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) Evaluation | At 12 weeks
  Wrinkle Severity Rating Scale (WSRS) evaluation at 12 weeks

SECONDARY OUTCOMES:
Wrinkle Severity Rating Scale (WSRS) Evaluation | At 2 weeks, 6 weeks
  Wrinkle Severity Rating Scale (WSRS) Evaluation at 2 weeks, and 6 weeks.
Global Aesthetic Improvement Scale (GAIS) Evaluation | At 2 weeks, 6 weeks and 12 weeks
  Global Aesthetic Improvement Scale (GAIS) Evaluation at 2 weeks, 6 weeks and 12 weeks.
VAS pain assessment at each time point | at injection and 15, 30, 45, and 60 min after injection
  VAS pain assessment at each time point (at injection and 15, 30, 45, and 60 min after injection)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seongnam-si, Gyeonggi-do
  - Chung-Ang University Hospital, Seoul